CLINICAL TRIAL: NCT04847401
Title: Evaluation of the Relationship Between Helicobacter Pylori Infection and Irritable Bowel Syndrome
Brief Title: the Relationship Between Helicobacter Pylori Infection and Irritable Bowel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reham Mohy El-Din Kamel, Resident doctor, Sohag University
Other Study IDs: Soh-Med-21-04-03
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Helicobacter Pylori; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: patients with Irritable Bowel Syndrome
  Interventions: Diagnostic Test: H. pylori stool antigen
- Group 2: normal
  Interventions: Diagnostic Test: H. pylori stool antigen

INTERVENTIONS:
Diagnostic Test: H. pylori stool antigen — using H. pylori antigen kits in stool

SUMMARY:
Evaluating any possible relationship between irritable bowel syndrome occurrence and Helicobacter pylori infection

ELIGIBILITY:
Inclusion Criteria:

* All patients will be selected according to Rome IV criteria for the diagnosis of IBS, which include:

Recurrent abdominal pain at least 1 day/week in the last 3 months, with two or more of the following criteria:

* Related to defecation
* Associated with a change in frequency of stool
* Associated with a change in form of stool. Criteria achieved for the last 3 months with symptom onset at least 6 months before diagnosis

Exclusion Criteria:

* • Rectal bleeding

  * Anemia
  * Weight loss
  * Onset after 50 years of age
  * Recent antibiotic use
  * Abnormal abdominal examination (organomegaly, lump)
  * Family history of colorectal cancer.
  * Family history of inflammatory bowel disease, or celiac disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: outpatient clinic patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-05-25 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
number of irritable bowel syndrome patients who had H.pylori infection | through study completion, an average of 1 year
  H.pylori stool antigen kits

IPD SHARING:
Plan to Share IPD: No